CLINICAL TRIAL: NCT01745159
Title: Proactive Treatment With Tacrolimus Ointment in Children With Moderate/Severe Atopic Dermatitis: A Randomized, Multicenter, Open-label Study
Brief Title: Preventive Treatment of Tacrolimus Ointment in Children With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACN-PRT-AD-12-1
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Moderate/Severe Atopic Dermatitis
Keywords: tacrolimus; Protopic; pediatric; atopic dermatitis; China
MeSH Terms: conditions — Lymphoma, Follicular; Dermatitis, Atopic | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- continued tacrolimus treatment (Experimental): children with moderate/severe atopic dermatitis treated with tacrolimus ointment and continuing to apply tacrolimus ointment during disease control period.
  Interventions: Drug: tacrolimus
- no additional treatment (No Intervention): children with moderate/severe atopic dermatitis treated with tacrolimus ointment and with no additional treatment during disease control period.

INTERVENTIONS:
Drug: tacrolimus
  Other Names: Protopic
  Arms: continued tacrolimus treatment

SUMMARY:
To assess if proactive, 2 times-weekly application of tacrolimus ointment can extend remission time to relapse and reduce the incidence of disease exacerbation (DE) in paediatric patients over a period of 6 months.

DETAILED DESCRIPTION:
This study includes three periods. First a screening period of up to one week. Second an open-label treatment period of up to six weeks where all participants apply tacrolimus ointment. Third an open-label disease control period of up to six months where half of the participants apply tacrolimus ointment and the other half of the participants do not apply treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as AD according to Williams diagnostic criteria.
2. Moderate or severe atopic dermatitis according to the criteria of Rajka and Langeland
3. At least approximately 10 % of body area
4. Patient is able to reach the centre within 3 days in case of a disease exacerbation.
5. Patient's legal representative(s) has/have given written informed consent. If the patient is capable of understanding the purposes and risks of the trial, written informed consent has been obtained from the patient as well

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Time to first DE (disease exacerbation) | 6 months of DCP(Disease Control Period) after 2 to 6 weeks of OLP(Open Label Period)

SECONDARY OUTCOMES:
Number of DEs during the DCP | 6 months of DCP (Disease Control Period)
Eczema Area and Severity Index (EASI) | 6 months of DCP (Disease Control Period) after 2 to 6 weeks of OLP (Open Label Period)
Investigator's Global Assessment (IGA) | 6 months of DCP (Disease Control Period) after 2 to 6 weeks of OLP (Open Label Period)
Duration of DE during DCP | 6 months of DCP (Disease Control Period)
The overall efficacy during OLP | After 2 to 6 weeks of OLP (Open Label Period)
Quantity of tacrolimus ointment used | 6 months of DCP (Disease Control Period) after 2 to 6 weeks of OLP (Open Label Period)
Incidence of adverse events | 6 months of DCP (Disease Control Period) after 2 to 6 weeks of OLP (Open Label Period)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (4):
- China (4):
  - Beijing
  - Chongqing
  - Guangzhou
  - Shanghai